CLINICAL TRIAL: NCT01261637
Title: Ultrasound Guided 0.25% Ropivacaine Transversus Abdominis Plane Block in Addition to Intrathecal Morphine and Multimodal Analgesia for the Management of Postoperative Pain Among Women Undergoing Cesarean Delivery.
Brief Title: Abdominal Wall Local Anesthesia to Maximize Postoperative Pain Control After Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Ronald George, Primary Investigator, MD, FRCPC, Assistant Professor, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IWK-4518-2009; IWK REB 4518
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Postoperative Pain
Keywords: cesarean, pain, transversus abdominus plane block
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.25% Ropivicaine (Experimental): 0.25% ropivicaine (maximum 1.5mg/kg)
  Interventions: Drug: Ropivicaine
- Placebo (Placebo Comparator): 20ml saline
  Interventions: Drug: Saline placebo

INTERVENTIONS:
Drug: Saline placebo — 20ml saline
  Arms: Placebo
Drug: Ropivicaine — 0.25% ropivicaine (maximum 1.5mg/kg)
  Other Names: Naropin
  Arms: 0.25% Ropivicaine

SUMMARY:
This study has been designed to determine if women undergoing cesarean delivery with spinal anesthesia and routine pain management who also have an additional ultrasound guided transversus abdominis plane (TAP)block using ropivacaine have better pain relief and a better quality of recovery than women who don't have the additional TAP block. Maximizing pain relief using ultrasound guided TAP blocks in addition to neuraxial opioids, NSAIDs, and acetaminophen may improve acute pain outcomes, reduce adverse side effects, and potentially reduce chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Non-emergent CD with planned spinal anesthesia
* American Society of Anesthesia physical status class I & II
* Age ≥ 18 years
* Term gestational age (≥ 37 weeks)
* English-speaking

Exclusion Criteria:

* Morbid Obesity (BMI³ 45 kg/m2)
* Laboring women
* Emergency CD
* Severe maternal cardiac disease
* Subjects with significant obstetric co-morbidities
* Failed spinal anesthesia
* Patient enrollment in another study involving medication within 30 days of CD
* Any other condition which may impair ability to cooperate with data collection
* Height less than 152 cm (5'0")
* Fetal anomalies or intrauterine fetal death

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be postoperative pain, measured by an NRS, the quality of recovery score (QoR) and a Self Assessment Diary in the first 24h postoperative period. | 24 hours

SECONDARY OUTCOMES:
NRS / QoR - 48 hour Opioid Consumption Side effects - nausea, sedation | 48 hours
TAP block success rates and duration of block effect will be assessed using a patient diary completed every 2 hours while the patient is awake. | 24 hours
Persistant pain outcomes will be assessed at 30 days and 6 months using 5-minute SF-36 health survey. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dolores McKeen, MD MSc FRCPC, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] McKeen DM, George RB, Boyd JC, Allen VM, Pink A. Transversus abdominis plane block does not improve early or late pain outcomes after Cesarean delivery: a randomized controlled trial. Can J Anaesth. 2014 Jul;61(7):631-40. doi: 10.1007/s12630-014-0162-5. Epub 2014 Apr 24. PMID 24764186